CLINICAL TRIAL: NCT01434628
Title: One Arm, Open Label, Prospective, Cohort Field Study to Assess the Safety and Efficacy of the PrePex Device for Non-Surgical Circumcision When Performed by Nurses in Resource Limited Settings for HIV Prevention
Brief Title: Cohort Field Study to Assess the Safety and Efficacy of the PrePex Device for Non-Surgical Circumcision When Performed by Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Vincent Mutabazi, Head of Reaserch RBC/IHDPC, Ministry of Health, Rwanda
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RMC-03
Record Dates: First submitted 2011-09-10; First posted 2011-09-15 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Male Circumcision; HIV Prevention
Keywords: Male Circumcision; HIV Prevention; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PrePex™ device (Experimental): Adult male circumcision by the PrePex™ device
  Interventions: Device: PrePex™ device

INTERVENTIONS:
Device: PrePex™ device — PrePex™ device for adult male circumcision. The PrePex™ device facilitates adult male circumcision that is bloodless with no anesthesia and no sutures

SUMMARY:
A range of observational and epidemiological studies have shown that the lifetime risk of HIV infection can be reduced by 70% through male circumcision.

Rwanda has a national plan to offer a voluntary male circumcision (MC) program to 2 million adult men in 2 years as part of a comprehensive HIV prevention strategy. To achieve this goal, the government launched a national study, based on the WHO Framework for Evaluation of Adult MC Devices, to assess the safety, efficacy and supremacy of the PrePex™ device when compared to surgical circumcision.

The PrePex device was developed to facilitate rapid scale up of non-surgical adult male circumcision in resource limited settings.

Rwanda validated the aforementioned endpoints via physicians in a Safety and Efficacy Study (NCT01150370) and Randomized, Controlled Comparison Study (NCT01284088). The procedure was bloodless, required no anesthesia, no sutures and no sterile settings, with 1 AE that was managed with minimal intervention.

Evidence submitted to members of WHO, USAID, UNAIDS and the Bill and Melinda Gates Foundation, and WHO audited the study site. The Safety and Efficacy study results were published in the JAIDS Journal of Acquired Immune Deficiency Syndromes, Sept 8, 2011, and presented in CROI 2011 and AUA 2011.

To achieve its national "catch up" campaign with minimal burden to the overly strained health system, which lacks physicians and surgical infrastructure, Rwanda needs to task shift the procedure to nurses. This study is meant to test the Safety and Efficacy in the hands of non-surgically trained nurses from the A1 and A2 cadres.

DETAILED DESCRIPTION:
Male circumcision can reduce the lifetime risk of HIV infection by 60% in high risk areas such as Sub Saharan Africa. In 2009, the US Government (USAID) reported that scaling up male circumcision to reach 80 percent of adult and newborn males in 14 African countries by 2015 could potentially avert more than 4 million adult HIV infections between 2009 and 2025 and yield annual cost savings of US$1.4 - 1.8 billion after 2015, with a total net savings of US$20.2 billion between 2009 and 2025.

There are over 38 million adolescent and adult males in Africa that could benefit from male circumcision for HIV prevention. The challenge Africa faces is how to safely scale up a surgical procedure in resource limited settings.

Rwanda has a national plan to offer a voluntary male circumcision (MC) program to 2 million adult men in 2 years as part of a comprehensive HIV prevention strategy. To achieve this goal, the government launched a national study, based on the WHO Framework for Evaluation of Adult MC Devices, to assess the safety, efficacy and supremacy of the PrePex™ device when compared to surgical circumcision.

The PrePex device was developed to facilitate rapid scale up of non-surgical adult male circumcision in resource limited settings.

Rwanda validated the aforementioned endpoints via physicians in a Safety and Efficacy Study (NCT01150370) and Randomized, Controlled Comparison Study (NCT01284088). The procedure was bloodless, required no anesthesia, no sutures and no sterile settings, with 1 AE that was managed with minimal intervention.

Evidence submitted to members of WHO, USAID, UNAIDS and the Bill and Melinda Gates Foundation, and WHO audited the study site. The Safety and Efficacy study results were published in the JAIDS Journal of Acquired Immune Deficiency Syndromes, Sept 8, 2011, and presented in CROI 2011 and AUA 2011.

To achieve its national "catch up" campaign with minimal burden to the overly strained health system, which lacks physicians and surgical infrastructure, Rwanda needs to task shift the procedure to nurses. This study is meant to test the Safety and Efficacy in the hands of non-surgically trained nurses from the A1 and A2 cadres.

The study will evaluate 75 subjects in training phase, 100 subjects in a pilot group and then additional 415 in a pivotal group summing up to 590.

The 503 subjects assigned to the Pivotal group will undergo standard PrePex procedure and follow up and will be the main core of the study. An interim safety report will be prepared after 100 subjects (Pilot Group). Up to 75 subjects will be enrolled to the Training group.

The study will assess the safety and efficacy of the PrePex device when circumcision is performed by nurses, among healthy adult men scheduled for voluntary circumcision, in preparation for scale up.

The Study duration per subject will be 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 - 54 years
* Subject wants to be circumcised
* Uncircumcised
* Able to understand the study procedures and requirements
* Agrees to abstain sexual intercourse and to keep caution not directly rub the cut area if masturbating, for 8 weeks.
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 7 weeks post removal (8 weeks total).
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
* Subject agrees to anonymous video and photographs of the procedure and follow up visits

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* Subject with the following diseases/conditions: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias,epispadias
* Known bleeding / coagulation abnormality, uncontrolled diabetes
* Subject who have an abnormal penile anatomy or any penile diseases
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits
* Refusal to take HIV test

Ages: 21 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 590 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the PrePex device when circumcision is performed by nurses | 8 weeks
  To assess the safety of the PrePex device by means of the following parameters: Clinical significant adverse event rate when circumcision is performed by nurses

SECONDARY OUTCOMES:
Evaluating the cost of PrePex circumcision procedure | 8 weeks
  Evaluating the cost of PrePex circumcision procedure when taking into account the following parameters:
  i. PrePex Procedure time and the resulting cost of provider's time
  ii. Cost of device training
  iii. Cost of staff time for follow-up visits
  iv. Cost of equipment and supplies needed for the circumcision procedure
To evaluate the PrePex training needs | 8 weeks
  Evaluation of the PrePex training needs and efficacy, including Direct measures by testing PrePex skills following participation in a formal training course Indirect measures of training efficacy by evaluating rate of AE and Average procedure time
Assessing ideal messaging for scale up sensitization, to include: | 8 weeks
  Assessing ideal messaging for scale up sensitization, to include:
  * Acceptability of the PrePex procedure by the patients and their partners
  * Indirect measures by collecting data on reasons to decline participation in the study and the percent of declining
  * Acceptability of the PrePex procedure by the care givers

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mutabazi, M.D., Principal Investigator — TRAC Plus
Locations (1):
- Kanombe Military Hospital, Kigali, Kigali, Rwanda